CLINICAL TRIAL: NCT06182982
Title: Efficacy of Auriculotherapy Medical Devices in Intraoperative Blood Pressure Control During Endoscopic Sinus Surgery, a Prospective Randomized Controlled Study.
Brief Title: Auriculotherapy for Intraoperative Blood Pressure Control
Acronym: AuriFESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID 5828
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Nasal Polyps; Anesthesia; Sinusitis; ENT Surgical Result - Nose Nasal Congestion
MeSH Terms: conditions — Nasal Polyps; Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricolotherapy (Experimental): Preoperative positioning of magnetic ball plasters for auricolotherpy.
  Interventions: Device: auricolotherapy
- Control (Sham Comparator): Ears will be covered by a band-aid (after a simulation of auricolotherapy)
  Interventions: Device: auricolotherapy

INTERVENTIONS:
Device: auricolotherapy — Magnetic bal plasters are applied on the ear surface

SUMMARY:
The endoscopic surgery of the paranasal sinuses (FESS) requires careful control of arterial pressure to prevent bleeding of the nasal mucosa that may lead to a reduction in the visual field. However, controlled reversible hypotension has been associated with phenomena of peripheral hypoperfusion with possible organ damage on an ischemic basis. Based on the data available in the literature, a mean arterial pressure (MAP) target between 50 and 65 mmHg is considered acceptable. Although blood pressure control is generally ensured through intravenous pharmacological approaches, there is evidence of efficacy with the use of Auriculotherapy medical devices (stimulation of specific points in the ear through the application of Magnetic ball plasters).

Proposed pharmacological choices to achieve this result have been multiple, although totally intravenous anesthesia with propofol and opioids seems to be more effective than balanced anesthesia with halogenated agents and opioids. However, this fundamental option requires the administration of antihypertensive drugs to achieve the blood pressure target. Despite common contraindications to individual pharmacological classes, various active principles have been compared. Among these, continuous low-dose nitroglycerin infusion has proven effective due to titratability linked to its short half-life, perioperative complications, and better conditions of peripheral perfusion compared to beta-blockers such as labetalol or esmolol.

Based on existing literature data, in our hospital, general anesthesia is typically conducted with intravenous techniques and the continuous administration of low doses of nitroglycerin in continuous infusion (0.01-2 mcg/kg/min). Despite the low dosages, this drug can be burdened with dosage-dependent adverse effects such as orthostatic hypotension, tachycardia, or headache. To reduce the dosage of nitroglycerin, we have borrowed from different contexts hypotensive auriculotherapy techniques (stimulation of specific ear points through the application of magnetic ball plasters), which have proven effective in managing systemic pressure in patients with essential hypertension.

These non-pharmacological techniques, already used during general anesthesia for the management of nausea and pain, could prove promising in reducing the use of antihypertensive drugs even in the intraoperative context. The primary hypothesis of our study is that the use of Auriculotherapy medical devices is effective in achieving a hypotensive effect in patients undergoing general anesthesia during FESS surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes to undergo Functional Endoscopic Sinus Surgery (FESS) under General Anesthesia
* Patients aged between 18 and 69 years
* History of well-controlled essential hypertension under pharmacological treatment for at least one year
* ASA Class II-III.

Exclusion Criteria:

* Age < 18 years;
* Pregnancy status;
* NYHA class > III;
* ASA class > III;
* BMI > 35;
* Positive history of Myocardial Infarction or neurovascular diseases;
* Previous treatment with antineoplastic agents;
* Secondary hypertension;
* Uncontrolled hypertension despite therapy (MAP > 125 in preoperative visit);
* Anatomic alterations of the auricles;
* Presence of carotid stenosis > 50%;
* Allergy or intolerance to drugs specified in the clinical protocol;
* Nickel or metal allergy present in magnetic spheres;
* Refusal of informed consent or inability to express it

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Nitroglycerin | at the end of surgery
  Reduction in the amount of intravenous nitroglycerin (mcg/kg/min) administered during FESS surgery

SECONDARY OUTCOMES:
Blood pressure | 24 hours
  Difference in blood pressure values between the two groups
Surgeon | at the end of surgery
  Subjective description by surgeon of the surgical field in terms of bleeding frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy